CLINICAL TRIAL: NCT02941263
Title: The Natural History of Geographic Atrophy Associated With Age-Related Macular Degeneration
Brief Title: Natural History of Geographic Atrophy Associated With Age-Related Macular Degeneration
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170008; 17-EI-0008
Record Dates: First submitted 2016-10-20; First posted 2016-10-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02-02

CONDITIONS: Age-Related Macular Degeneration
Keywords: Eye Disease; Natural History
MeSH Terms: conditions — Macular Degeneration; Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected Participants: Participants with unilateral or bilateral GA associated with atrophic AMD.

SUMMARY:
Background:

Age-related macular degeneration (AMD) affects the macula in the eye. This is the central part of the retina. It is needed for sharp, clear vision and activities like reading and driving. AMD is the leading cause of vision loss in Americans 60 years of age and older. An advanced form of AMD is called geographic atrophy or GA. It happens when light-sensitive cells in the macula die so much that central vision decreases.

Objective:

To learn more about geographic atrophy associated with age-related macular degeneration.

Eligibility:

Adults at least 55 years old with a certain kind of GA. They must be enrolled in study 08-EI-0102, 08-EI-0169, 08-EI-0043, 12-EI-0042, or 11-EI-0147 but no other studies.

Design:

Participants will be screened with medical history, physical exam, and an eye exam.

Participants will have study visits every 3 months for 15 months, then every 6 months. They will be in the study almost 4 years.

Visits will last about 8 hours. At each visit, participants may have:

* Medical and eye history. Participants will answer questions about their general health and eye health. They may answer written questions about how their eye problems affect their life.
* Eye exam and photographs. Eye pressure will be measured and eye movements will be checked. Pupils will be dilated with drops. The thickness of the retina will be measured and photos of the eye may be taken.

DETAILED DESCRIPTION:
Objective: Age-related macular degeneration (AMD), the leading cause of blindness in people over age 65 in the United States, is a heterogeneous clinical entity in which retinal degeneration occurs predominantly in the macula in the context of aging and leads to impairment of central visual acuity (VA). AMD occurs in two general forms, one of which involves choroidal neovascularization (CNV) with subsequent formation of a disciform scar. This is often referred to as the neovascular or wet form. A second form, the subject of this study, is termed dry atrophic macular degeneration or otherwise geographic atrophy (GA) and involves a slow progressive atrophy of retinal pigment epithelial (RPE) cells and photoreceptors in the macula, also resulting in central vision loss. GA is estimated to affect up to one million people in the U.S. and there is no current treatment that can prevent its onset. While the etiology of GA is not completely understood, inflammatory processes involving the activation of resident immune cells of the retina called microglia are likely to contribute. The objective of this study is to study the progression of GA so as to be able to characterize in quantitative terms the natural progression of GA in patients, whether or not they are receiving any directed treatment.

Study Population: Twenty-five (25) participants with unilateral or bilateral GA associated with AMD will be enrolled.

Design: This prospective, natural history study will follow participants with GA associated with AMD.

Outcome Measures:

The primary outcome is the rate of change in area of GA based on grading by an external Reading Center of fundus autofluorescence (FAF) images in the assigned study eye. The primary outcome will be calculated for 45 months as compared to baseline.

Secondary outcomes will include changes in best-corrected visual acuity (BCVA), rate of change in area of GA based on fundus photography and development of exudative AMD ascertained using optical coherence tomography (OCT) and changes in macular sensitivity.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible, the following inclusion criteria must be met, where applicable.

1. Participant must be 55 years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant must have evidence of early or intermediate AMD as defined by characteristic presence of drusen and/or pigmentary changes.
4. Participant is enrolled in one of the following screening protocols: 08-EI-0102, 08-EI-0169 (closed), 08-EI-0043, 12-EI-0042, 11-EI-0147, or 16-EI-0134.

EXCLUSION CRITERIA:

A participant is not eligible if any of the following exclusion criteria are present.

1. Participant is actively receiving study therapy in another investigational study.
2. Participant is unable to comply with study procedures or follow-up visits.
3. Participant is on ocular or systemic medications known to be toxic to the lens, retina or optic nerve (e.g., ethambutol, chloroquine, or hydroxychloroquine).

STUDY EYE ELIGIBILITY CRITERIA:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

STUDY EYE INCLUSION CRITERIA:

1. The study eye(s) must have GA compatible with dry AMD. GA is defined as one or more well-defined and often circular patches of partial or complete depigmentation of the RPE, typically with exposure of underlying choroidal blood vessels. Even if much of the RPE appears to be preserved and large choroidal vessels are not visible, a round patch of RPE partial depigmentation may be classified as early GA. The GA in the study eye must be able to be photographed in their entirety and it must not be contiguous with any areas of peripapillary atrophy, which can complicate area measurements.
2. The study eye(s) must have clarity of ocular media and degree of pupil dilation sufficient to permit adequate fundus photographs.

STUDY EYE EXCLUSION CRITERIA:

1. Current evidence of neovascularization as determined by the treating physician or a history of treatments for neovascularization.
2. Evidence of retinal atrophy due to causes other than atrophic AMD.
3. Current evidence or history of ocular disorders in the study eye that might confound study outcome measures, including (but not limited to):

   1. non-proliferative diabetic retinopathy involving 10 or more hemorrhages or microaneurysms, or active proliferative diabetic retinopathy
   2. Branch or central retinal vein or artery occlusion
   3. Macular hole
   4. Pathologic myopia
   5. Uveitis
   6. Pseudovitelliform maculopathy
4. History of vitreoretinal surgery.
5. Need for ocular surgery during the course of the study.
6. Recent history of lens removal (< 3 months prior to enrollment) or Yttrium Aluminum Garnet (YAG) laser capsulotomy (< 1 month prior to enrollment).

Ages: 55 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-five (25) participants, age 55 years and older, with unilateral or bilateral GA associated with atrophic AMD will be accrued.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the difference in the mean rate of change in area of GA in the study eye based on digital grading of FAF images by an external Reading Center. | Calculated 45 months as compared to baseline
  Difference in the mean rate of change in area of GA in the study eye based on digital grading of FAF images by an external Reading Center.

SECONDARY OUTCOMES:
Differences in study eyes for the following: mean rate of change in area of GA based on digital grading of color fundus images, mean changes in BCVA, mean changes in central retinal thickness on OCT, and the proportion of study eyes developing w... | 45 months as compared to baseline
  Differences in the study eyes for the following outcome measures: mean rate of change in area of GA based on digital grading of color fundus images by an external reading center, mean changes in BCVA, mean changes in central retina thickness on OCT and the proportion of study eyes developing wet AMD determined by OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Tiarnan DL Keenan, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2017-EI-0008.html